CLINICAL TRIAL: NCT00765986
Title: A Study to See if a New Type of Imaging Can Help Our Understanding of the Course of Non-small Cell Lung Cancer in Patients Undergoing Treatment With Radiotherapy or Chemoradiotherapy
Brief Title: Pilot Study of 18F-FAZA in Assessing Early Functional Response in Patients With Inoperable Non Small Cell Lung Cancer Undergoing Radiotherapy or Chemo-radiotherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: LU-24319
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2014-10

CONDITIONS: Lung Neoplasm; Cell Hypoxia
Keywords: 18F-FAZA; 18F-FDG; Positron Emission Tomography
MeSH Terms: conditions — Lung Neoplasms | interventions — fluoroazomycin arabinoside; Fluorodeoxyglucose F18

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with inoperable NSCLC undergoing RT or Chemo-RT
  Interventions: Other: 18F-FAZA; Other: 18F-Fluorodeoxyglucose (18F-FDG)

INTERVENTIONS:
Other: 18F-FAZA — Radioactive dose of 110-600 MBq per injection. Up to a maximum of 6 injections per patient: pre-Tx, after 4 weeks (20 fractions) of RT, then 4 weeks, 90 days and 12 months post-RT and upon logo-regional progression or recurrence.
  Other Names: NAP
Other: 18F-Fluorodeoxyglucose (18F-FDG) — Radioactive dose of 100-710 MBq per injection. Up to a maximum of 6 injections per patient: pre-Tx, after 4 weeks (20 fractions) RT, then 4 weeks, 90 days, and 12 months post-RT, and upon loco-regional progression or recurrence.
  Other Names: FluGlucoScan Injection

SUMMARY:
Non-small cell lung cancer (NSCLC) has a poor prognosis if not caught early enough. One of the factors that may impact the ability to control NSCLC is low oxygen levels (hypoxia) inside the tumour. This study will use 18F-FAZA PET scans to assess whether patients have hypoxic tumours and to monitor the changes to the hypoxic areas of a tumour during currently available standard treatment. It is hypothesized that 18F-FAZA PET may predict response to treatment, local control, and/or survival in NSCLC.

DETAILED DESCRIPTION:
Locally advanced NSCLC has a poor prognosis with a 5 year overall survival rate of only 15%. Tumour hypoxia may impact the ability to control NSCLC. Using 18F-FAZA PET, this study will assess patients for hypoxic treatment. With this information, we can start individualizing patient treatment to target hypoxia. The relationship between areas of hypoxia (18F-FAZA) and high glucose utilization (18F-FDG) will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically-proven, by biopsy or cytology, unresected lung cancer of the following histological types: squamous cell carcinoma; adenocarcinoma; undifferentiated large cell carcinoma, and non-small cell, not otherwise specified (NOS, diagnosis on cytology alone)
2. Patients with American Joint Committee on Cancer (AJCC) Stage I, II, IIIA, or IIIB with detectable tumour that can be encompassed by radiation therapy fields, including both primary tumour and the involved regional lymph nodes.
3. Patients must be deemed to be suitable to undergo definitive (i.e. potentially curable) chemoradiotherapy or radiotherapy by the treating Physician.
4. The prescribed radiotherapy dose must be a minimum of 60 Gy in 30 fractions
5. Male or female ≥ 18 years of age. If female of child bearing potential and outside the window of 10 days since the first day of the last menstrual period, a negative pregnancy test is required.
6. ECOG/Zubrod status 0-1
7. Patients must have at least one measurable lesion ≥ 1 cm on CT
8. Able and willing to follow instructions and comply with the protocol
9. Provide written informed consent prior to participation in the study

Exclusion Criteria:

1. Patients who have undergone complete or subtotal tumour resection
2. Patients with post-resection intrathoracic tumour recurrence
3. Patients eligible for definitive surgery (patients who are eligible for surgery, but surgery did not proceed are eligible for this trial)
4. No distant or metastasis, prior chemotherapy, or thoracic neck or radiotherapy
5. Evidence of any small cell histology
6. Prior or concurrent malignancy (except non-melanomatous skin cancer) unless disease-free for at least 5 years
7. Inability to lay in supine position for approximately one hour
8. Nursing or pregnant females
9. Aged less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with inoperable NSCLC undergoing radiotherapy or chemoradiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2008-10; Primary Completion 2015-09 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
To determine the relationship between hypoxic changes and the early local tumour response after definitive radiotherapy or chemoradiotherapy in NSCLC | 2.5 yrs

SECONDARY OUTCOMES:
To establish if a correlation exists between 18F-FAZA PET and FluGlucoScan Injection PET in determining responses to definitive treatment in NSCLC | 2.5 yrs
To assess if patterns of local failure/overall survival correlate with 18F-FAZA PET and/or FluGlucoScan Injection PET | 7 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Wilson Roa, MD, Principal Investigator — wilson.roa@albertahealthservices.ca
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada